CLINICAL TRIAL: NCT05013151
Title: The Effect of Dates and Castor Oil on the Initiation of Spontaneous Labor in Primigravida Parturients- a Prospective Randomized Trial
Brief Title: The Effect of Dates and Castor Oil on the Initiation of Spontaneous Labor in Primigravida Parturients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Nir Kugelman, Dr. Nir Kugelman, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-21-0064-CTIL
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Effect of Dates and Castor Oil on Spontaneous Labor
MeSH Terms: interventions — Chronology as Topic; Castor Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Date consumption (Experimental): Consumption of 6 dates a day until 41 weeks of gestation
  Interventions: Dietary Supplement: Dates
- Castor oil consumption (Experimental): One time consumption of 60 CC of Castor oil
  Interventions: Dietary Supplement: Castor oil
- Control Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Dates — Consumption of 6 dates a days until 41 weeks of gestation
  Arms: Date consumption
Dietary Supplement: Castor oil — One time consumption of 60 CC Castor oil
  Arms: Castor oil consumption

SUMMARY:
Finding a natural and efficient method to improve the chance of entering spontaneous labor beyond 39 weeks of gestation will address both the medical necessity and the will of many parturients to avoid medical interventions.

In this study we aim to evaluate the effect of dates and castor oil on the initiation of spontaneous labor in primigravida parturients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who come to the obstetrical emergency department for normal check up between 39+4 and 40+2 weeks of gestation
* Primipara
* Bishop cervical score below 5
* Low risk pregnancy
* Singleton pregnancy
* Vertex presentation
* Women who haven't consumed dates over once a week in month prior the checkup and haven't consumed castor oil prior to enrollment.

Exclusion Criteria:

* Any medical indication for labor induction
* Regular contractions
* Premature rupture of membranes
* Women who consumed dates over once a week in month prior the checkup or consumed castor oil prior to enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-08-24 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Rates of spontaneous entry into labor | 2 weeks after enrollment
  Rate of women who will enter labor spontaneously without intervention

SECONDARY OUTCOMES:
Cervical ripening- Bishop score | 2 weeks after enrollment
  Change of cervical ripening status after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lena Sagi-Dain, MD, Study Director — Lady Davis Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No